CLINICAL TRIAL: NCT06610292
Title: Effects of Pharmacist-led Medication Reconciliation Services on Geriatric Patients At a Leading Military Hospital in Jordan
Brief Title: Effects of Pharmacist-led Medication Reconciliation Services on Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Jordanian Royal Medical Services (Other); Royal Medical Services, Jordanian Armed Forces (Other)
Responsible Party: Principal Investigator, Majed Shafaamri, Research Assistant, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6/2018
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Geriatric Patients; Medication Reconcilitation Upon Hospital Admission; Medication Reconciliation At Discharge; Pharmacist-led Medication Reconciliation
Keywords: Medication reconciliation; Geriatrics; Geriatric patients; Jordan; Tertiary military hospital; Pharmacist-led medication reconciliation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients did not receive Pharmacist-led medication reconciliation services
- Intervention group (Experimental): Patients received Pharmacist-led medication reconciliation services
  Interventions: Other: Pharmacist-led medication reconciliation services

INTERVENTIONS:
Other: Pharmacist-led medication reconciliation services — Upon admission, information about patients Best Possible Medication History (BPMH) was extracted. Information on current medications, both regular and as-needed, was also recorded. All data were cross-referenced with the electronic records and verified through patients or caregivers interviews to create a comprehensive medication list.
  Then, comparison was conducted between standard care medication list and Pharmacist-led medication reconciliation list to identify any possible medication discrepancies. Also, during hospital stay and upon discharge emerging medication discrepancies were assessed and resolved.
  Moreover, the impacts on healthcare resources utilization within 30 days post-discharge was measured. This includes evaluating hospital re-admissions, emergency department visits, and the occurrence of any adverse drug events (ADEs).
  Arms: Intervention group

SUMMARY:
This study aims to assess the effects of Pharmacist-led medication reconciliation on hospitalized elderly patients aged above 65 at a leading tertiary military hospital in Jordan.

DETAILED DESCRIPTION:
A four-month randomized controlled trial was conducted at King Hussein Medical Hospital (KHMH), one of the Royal Military Medical Services (RMS) tertiary hospitals located in central Amman. During the study period, 128 patients were selected using convenience sampling. Later, medication histories were compared between pre-admission and admission records to obtain the Best Possible Medication History (BPMH) and identify medication discrepancies, which were categorized as either intentional (documentation errors) or unintentional discrepancies.

The already selected patients were randomly allocated into two groups (intervention and control groups). Then, Pharmacist-led medication reconciliation services were provided to the intervention group and standard care was provided to the control group. Also at discharge the number of medication discrepancies was documented. Linear regression analysis was performed to assess risk factors associated with the occurrence of unintentional discrepancies.

Within 30 days post-discharge, patients were assessed for any hospital re-admissions, emergency department visits and medication-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patient within no more than 24 hours and anticipated to stay in the hospital for more than 48 hours.
* Geriatrics patients defined as those aged (≥65 years) (Orimo et al., 2006).
* Prescribed at least one chronic medication prior to the study admission.

Exclusion Criteria:

* Patient admitted to the critical care or isolation units or in unconscious or comatose states.
* Patients if they were discharged against medical advice.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Describing prevalence and nature of medication discrepancies in elderly patients and investigating contributing factors to medication discrepancies. | Up to 20 weeks
  Linear regression analysis was performed to assess risk factors associated with the occurrence of medication discrepancies in elderly patients.
Analysis of the effects of Pharmacist-led medication reconciliation services on resolving medication discrepancies upon discharge | Up to 16 weeks
  Number of resolved medication discrepancies was documented upon discharge after providing pharmacist-led medication reconciliation services.
Evaluating the impacts of Pharmacist-led medication reconciliation services on hospital re-admissions within 30 days of discharge | Up to 20 weeks
  Elderly patients were assessed for number of hospital re-admissions within 30 days of discharge at control and intervention groups.
Evaluating the impacts of Pharmacist-led medication reconciliation services on emergency department visits within 30 days of discharge | Up to 20 weeks
  Elderly patients were assessed for number of emergency department visits within 30 days of discharge at control and intervention groups.
Evaluating the impacts of Pharmacist-led medication reconciliation services on medications side effects within 30 days of discharge | Up to 20 weeks
  Elderly patients were assessed for incidence of medications side effects within 30 days of discharge at control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Hammad, Principal Investigator — Department of Biopharmaceutics and Clinical Pharmacy, School of Pharmacy, University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No